CLINICAL TRIAL: NCT00725738
Title: Intracoronary Autologous Stem Cell Transplantation in ST Elevation Myocardial Infarction: TRACIA Study.
Acronym: TRACIA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Heart Institute, Mexico (Other Government)
Collaborators: National Center of Blood Transfusion Mexico. (Unknown)
Responsible Party: Marco Antonio Peña Duque MD Interventional Cardiologist, National Institute of Cardiology "Ignacio Chávez"
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-583
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2008-07

CONDITIONS: Acute Myocardial Infarction
Keywords: Myocardial; Infarction,; Stem; Cell; Therapy
MeSH Terms: conditions — Infarction | interventions — Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Stem Cell Transplantation Group: Between the fifth and seventh day post-primary angioplasty (PTCA) we extract the stem cell from iliac crest and during the same day the patient undergoes to a new cardiac catheterization in which we perform the intracoronary injection (about 1-2 million of CD34 cells) through the infarct related artery by a PTCA "over-the-wire" catheter.
  Interventions: Genetic: Stem Cell Transplantation

INTERVENTIONS:
Genetic: Stem Cell Transplantation — 1-2 million of CD34 cells injected through the infarct related artery by PTCA "over-the-wire" catheter during multiple sequences of balloon artery occlusion with a mean duration of 30 minutes.
  Other Names: Stem Cell

SUMMARY:
The purpose of this study is to evaluate the ejection fraction (EF) increase at 6 months follow up and major adverse cardiovascular events (MACE) after intracoronary autologous stem cell transplantation in ST elevation myocardial infarction patients versus a control group.

DETAILED DESCRIPTION:
Experimental trials with bone marrow cell have suggested that adult stem cell can contribute to regeneration of infarcted myocardial muscle and increase the neovascularization of the ischemic tissue.

Post-myocardial infarction heart failure secondary to ventricular remodelation it's an increasing problem. A novel therapeutic approach for decrease this consequence is to induce the angiogeneses and regeneration of myocardial cells.

Many trials have shown benefits through the intracoronary injection of stem cell, however the clinical benefit is still controversial. The present trial is a randomized single blinded controlled trial designed to evaluate the improvement on EF and survival in post ST elevation myocardial infarction patients undergoing to intracoronary autologous stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Both gender patients between 20 and 75 years old with an acute myocardial infarction (less 24 hrs of symptoms) undergoing to primary angioplasty.
* LVEF < o = 45% by MRI, radioisotopic ventriculography or echocardiogram.
* Informed written consent.

Exclusion Criteria:

* Cardiogenic Shock.
* Post-myocardial infarction mechanical complication
* Malignant ventricular arrythmias
* History of malignant disease during the last five years.
* Pregnancy
* Renal chronic disease with a creatinine level > 2.6 mg/dl.
* Any kind of stroke during the last year.
* Any chronic disease that can affect the patient survival during the trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the mean LVEF increase by magnetic resonance imaging (MRI) at 6 months of follow up between the stem cell group and the control group. | 6 months

SECONDARY OUTCOMES:
Evaluate the left ventricular end diastolic volume (LVEDV) and left ventricular end systolic volume (LVESV)with image magnetic resonance(IMR) at 6 months follow up between stem cell and control group. | 6 months
Evaluate the oxygen consumption during treadmill stress test (MVO2) by expired gases analysis and the incidence of MACE at 6 months follow up between stem cell and control group. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marco A Peña-Duque, MD, Principal Investigator — National Institute of Cardiology "Ignacio Chávez" Mexico; Marco A Peña-Duque, MD, Study Director — National Institute of Cardiology "Ignacio Chávez" Mexico; Marco A Peña-Duque, MD, Study Chair — National Institute of Cardiology "Ignacio Chávez" Mexico
Locations (1):
- National Institute of Cardiology "Ignacio Chávez" Mexico, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Lange RA, Hillis LD. Reperfusion therapy in acute myocardial infarction. N Engl J Med. 2002 Mar 28;346(13):954-5. doi: 10.1056/NEJM200203283461302. No abstract available. PMID 11919303
- [Background] Keeley EC, Boura JA, Grines CL. Primary angioplasty versus intravenous thrombolytic therapy for acute myocardial infarction: a quantitative review of 23 randomised trials. Lancet. 2003 Jan 4;361(9351):13-20. doi: 10.1016/S0140-6736(03)12113-7. PMID 12517460
- [Background] Giugliano RP, Braunwald E; TIMI Study Group. Selecting the best reperfusion strategy in ST-elevation myocardial infarction: it's all a matter of time. Circulation. 2003 Dec 9;108(23):2828-30. doi: 10.1161/01.CIR.0000106684.71725.98. No abstract available. PMID 14662688
- [Background] Pitt B, Remme W, Zannad F, Neaton J, Martinez F, Roniker B, Bittman R, Hurley S, Kleiman J, Gatlin M; Eplerenone Post-Acute Myocardial Infarction Heart Failure Efficacy and Survival Study Investigators. Eplerenone, a selective aldosterone blocker, in patients with left ventricular dysfunction after myocardial infarction. N Engl J Med. 2003 Apr 3;348(14):1309-21. doi: 10.1056/NEJMoa030207. Epub 2003 Mar 31. PMID 12668699
- [Background] Pfeffer MA, McMurray JJ, Velazquez EJ, Rouleau JL, Kober L, Maggioni AP, Solomon SD, Swedberg K, Van de Werf F, White H, Leimberger JD, Henis M, Edwards S, Zelenkofske S, Sellers MA, Califf RM; Valsartan in Acute Myocardial Infarction Trial Investigators. Valsartan, captopril, or both in myocardial infarction complicated by heart failure, left ventricular dysfunction, or both. N Engl J Med. 2003 Nov 13;349(20):1893-906. doi: 10.1056/NEJMoa032292. Epub 2003 Nov 10. PMID 14610160
- [Background] Orlic D, Kajstura J, Chimenti S, Jakoniuk I, Anderson SM, Li B, Pickel J, McKay R, Nadal-Ginard B, Bodine DM, Leri A, Anversa P. Bone marrow cells regenerate infarcted myocardium. Nature. 2001 Apr 5;410(6829):701-5. doi: 10.1038/35070587. PMID 11287958
- [Background] Kocher AA, Schuster MD, Szabolcs MJ, Takuma S, Burkhoff D, Wang J, Homma S, Edwards NM, Itescu S. Neovascularization of ischemic myocardium by human bone-marrow-derived angioblasts prevents cardiomyocyte apoptosis, reduces remodeling and improves cardiac function. Nat Med. 2001 Apr;7(4):430-6. doi: 10.1038/86498. PMID 11283669
- [Background] Strauer BE, Brehm M, Zeus T, Kostering M, Hernandez A, Sorg RV, Kogler G, Wernet P. Repair of infarcted myocardium by autologous intracoronary mononuclear bone marrow cell transplantation in humans. Circulation. 2002 Oct 8;106(15):1913-8. doi: 10.1161/01.cir.0000034046.87607.1c. PMID 12370212
- [Background] Wollert KC, Meyer GP, Lotz J, Ringes-Lichtenberg S, Lippolt P, Breidenbach C, Fichtner S, Korte T, Hornig B, Messinger D, Arseniev L, Hertenstein B, Ganser A, Drexler H. Intracoronary autologous bone-marrow cell transfer after myocardial infarction: the BOOST randomised controlled clinical trial. Lancet. 2004 Jul 10-16;364(9429):141-8. doi: 10.1016/S0140-6736(04)16626-9. PMID 15246726
- [Background] Fernandez-Aviles F, San Roman JA, Garcia-Frade J, Fernandez ME, Penarrubia MJ, de la Fuente L, Gomez-Bueno M, Cantalapiedra A, Fernandez J, Gutierrez O, Sanchez PL, Hernandez C, Sanz R, Garcia-Sancho J, Sanchez A. Experimental and clinical regenerative capability of human bone marrow cells after myocardial infarction. Circ Res. 2004 Oct 1;95(7):742-8. doi: 10.1161/01.RES.0000144798.54040.ed. Epub 2004 Sep 9. PMID 15358665
- [Background] Schachinger V, Erbs S, Elsasser A, Haberbosch W, Hambrecht R, Holschermann H, Yu J, Corti R, Mathey DG, Hamm CW, Suselbeck T, Assmus B, Tonn T, Dimmeler S, Zeiher AM; REPAIR-AMI Investigators. Intracoronary bone marrow-derived progenitor cells in acute myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1210-21. doi: 10.1056/NEJMoa060186. PMID 16990384
- [Background] Lunde K, Solheim S, Aakhus S, Arnesen H, Abdelnoor M, Egeland T, Endresen K, Ilebekk A, Mangschau A, Fjeld JG, Smith HJ, Taraldsrud E, Grogaard HK, Bjornerheim R, Brekke M, Muller C, Hopp E, Ragnarsson A, Brinchmann JE, Forfang K. Intracoronary injection of mononuclear bone marrow cells in acute myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1199-209. doi: 10.1056/NEJMoa055706. PMID 16990383
- [Background] Abdel-Latif A, Bolli R, Tleyjeh IM, Montori VM, Perin EC, Hornung CA, Zuba-Surma EK, Al-Mallah M, Dawn B. Adult bone marrow-derived cells for cardiac repair: a systematic review and meta-analysis. Arch Intern Med. 2007 May 28;167(10):989-97. doi: 10.1001/archinte.167.10.989. PMID 17533201
- [Background] Assmus B, Honold J, Schachinger V, Britten MB, Fischer-Rasokat U, Lehmann R, Teupe C, Pistorius K, Martin H, Abolmaali ND, Tonn T, Dimmeler S, Zeiher AM. Transcoronary transplantation of progenitor cells after myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1222-32. doi: 10.1056/NEJMoa051779. PMID 16990385
- [Background] Myers J, Prakash M, Froelicher V, Do D, Partington S, Atwood JE. Exercise capacity and mortality among men referred for exercise testing. N Engl J Med. 2002 Mar 14;346(11):793-801. doi: 10.1056/NEJMoa011858. PMID 11893790
- [Background] Gibbons RJ, Balady GJ, Bricker JT, Chaitman BR, Fletcher GF, Froelicher VF, Mark DB, McCallister BD, Mooss AN, O'Reilly MG, Winters WL, Gibbons RJ, Antman EM, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Russell RO, Smith SC; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Committee to Update the 1997 Exercise Testing Guidelines. ACC/AHA 2002 guideline update for exercise testing: summary article. A report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee to Update the 1997 Exercise Testing Guidelines). J Am Coll Cardiol. 2002 Oct 16;40(8):1531-40. doi: 10.1016/s0735-1097(02)02164-2. No abstract available. PMID 12392846
- [Background] Sutton MG, Sharpe N. Left ventricular remodeling after myocardial infarction: pathophysiology and therapy. Circulation. 2000 Jun 27;101(25):2981-8. doi: 10.1161/01.cir.101.25.2981. No abstract available. PMID 10869273
- [Background] Froelicher V, Myers J. Exercise and the heart. Fourth edition. Ed. Saunders. Philadelphia 2000. pp 456.